CLINICAL TRIAL: NCT06073483
Title: Exploratory Study of Toumai Endoscopic Surgery System for Remote Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE-04
Record Dates: First submitted 2023-09-07; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5G remote gastrectomy (Experimental)
  Interventions: Device: Toumai Endoscopic surgery System

INTERVENTIONS:
Device: Toumai Endoscopic surgery System — 5G remote gastrectomy on subjects using the Toumai endoscopic surgery system

SUMMARY:
This clinical study was a prospective, single-center, single-arm exploratory study. Subjects who meet the inclusion criteria will be enrolled in this study, where surgeons will perform 5G remote gastrectomy on subjects using the Toumai endoscopic surgery system, and explore and evaluate the safety and efficacy of this clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ actual age ≤80 years old.
2. Patients requiring gastrointestinal endoscopic surgery.
3. Willing to cooperate with and complete the study follow-up and related examinations.
4. Voluntarily participate in the study and sign the informed consent in person.

Exclusion Criteria:

1. Have serious cardiovascular or circulatory disease and cannot tolerate surgery.
2. Participated in other clinical trials within the last 3 months.
3. Inability to understand trial requirements, or inability to complete the study follow-up plan.
4. Researchers believe that there are other circumstances that are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The rate of intraoperative complications | The day of surgery
  Intraoperative complications, including organ injury and vascular injury, were evaluated using the Satava grading system to determine whether the occurrence of complications was related to the study instrument or surgery
The rate of postoperative complications | Postoperative 30 days
  Postoperative complications, including postoperative bleeding, fever, and incisional infection, were evaluated using the Clavien-Dindo grading system to determine whether the occurrence of complications was related to the study instrument or surgery.

SECONDARY OUTCOMES:
Intraoperative system failure rate | The day of surgery
Surgical completion rate | The day of surgery
Intraoperative blood loss | The day of surgery
Operation time | The day of surgery
Preoperative device assembly time | The day of surgery
Intraoperative instrument operation error rate | The day of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China